CLINICAL TRIAL: NCT04809376
Title: A 2-stage, Adaptive, Randomised, Double-blind, Placebo-controlled, Multicentre Study to Evaluate Dose and Treatment Effect of Pentosan Polysulfate Sodium Compared With Placebo in Participants With Knee Osteoarthritis Pain
Brief Title: Treatment Effects of Subcutaneous Injections of Pentosan Polysulfate Sodium vs Placebo in Participants With Knee OA Pain
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Paradigm Biopharmaceuticals USA (INC) (Industry)
Responsible Party: Sponsor
Organization: Paradigm Biopharmaceuticals Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARA_OA_002
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride; Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PPS Twice Weekly (Experimental): Pentosan Polysulfate Sodium (PPS) twice weekly for 6 weeks
  Interventions: Drug: Pentosan Polysulfate Sodium twice weekly
- PPS Once Weekly (Experimental): Pentosan Polysulfate Sodium (PPS) + placebo once weekly for 6 weeks
  Interventions: Drug: Placebo (Sodium Chloride Injection, 0.9%); Drug: Pentosan Polysulfate Sodium once weekly
- PPS Fixed Dose Once Weekly (Experimental): Pentosan Polysulfate Sodium (PPS) Fixed dose (100mg,150mg, or 180mg) once weekly + placebo once weekly for 6 weeks
  Interventions: Drug: Placebo (Sodium Chloride Injection, 0.9%); Drug: Pentosan Polysulfate Sodium Fixed Dose
- Placebo (Placebo Comparator): Placebo twice weekly for 6 weeks
  Interventions: Drug: Placebo (Sodium Chloride Injection, 0.9%)

INTERVENTIONS:
Drug: Pentosan Polysulfate Sodium twice weekly — Subcutaneous Injection, 1.5mg/kg Ideal body Weight (IBW)
  Other Names: PPS twice weekly
  Arms: PPS Twice Weekly
Drug: Placebo (Sodium Chloride Injection, 0.9%) — Placebo to match PPS
  Other Names: Placebo
  Arms: PPS Fixed Dose Once Weekly; PPS Once Weekly; Placebo
Drug: Pentosan Polysulfate Sodium Fixed Dose — Subcutaneous Injection, 100/150/180 mg if <65kg/ ≥ 65 kg and ≤ 90kg/ >90 kg IBW
  Other Names: Fixed Dose
  Arms: PPS Fixed Dose Once Weekly
Drug: Pentosan Polysulfate Sodium once weekly — Subcutaneous Injection, 2.0mg/kg Ideal body Weight (IBW)
  Other Names: PPS once weekly
  Arms: PPS Once Weekly

SUMMARY:
The purpose of this study is to measure the change in pain and function with subcutaneous injections of pentosan polysulfate sodium (PPS) compared with subcutaneous injections of placebo in participants with knee osteoarthritis pain.

Study details include:

* The study duration will be up to 31 weeks per participant
* The treatment duration will be 6 weeks.
* The visit frequency will be twice weekly during treatment.
* The visit frequency will be every 4 weeks during the follow-up period.

DETAILED DESCRIPTION:
This is a 2-stage, adaptive, randomized, double-blind, placebo-controlled, multicenter study that will evaluate the dose and treatment effect of PPS in participants with knee OA pain.

In Stage 1 (dose selection), approximately 468 participants will be randomised 1:1:1:1 to receive 1 of 3 PPS dose regimens or placebo for 6 weeks. A minimum of 96 participants (24 within each dose group) will be assigned to the Pharmacokinetic (PK) subset.

Participants in Stage 1 will be randomly allocated to receive:

* 1.5 mg/kg calculated for ideal body weight (IBW) PPS twice weekly
* 2 mg/kg IBW PPS once weekly + placebo once weekly
* 100/150/180 mg PPS if ≤ 65 kg/ ≥ 65 kg and ≤ 90kg/ > 90kg IBW+ placebo once weekly
* placebo twice weekly

In Stage 2, approximately 470 participants will be randomized 1:1 to receive the selected PPS dose regimen or placebo for 6 weeks. Approximately 150 participants (75 per group) will be assigned to the PK subset.

Participants in Stage 2 will be randomly allocated to receive:

* One of the 3 Stage 1 PPS dose regimens selected by the DMC
* placebo twice weekly

The maximum duration for each participant is approximately 31 weeks, which includes:

* 7-week Screening Period from Day -45 to Day -1
* 6-week Treatment Period from Day 1 to Day 39
* 18-week Follow-up Period from Day 40 to Day 168

ELIGIBILITY:
Inclusion Criteria:

* Participant must be >= 18 years of age inclusive, at the time of signing the informed consent.
* Clinical diagnosis of OA in the index knee by American College of Rheumatology criteria 1986 criteria.
* Radiographic diagnosis (confirmed by radiologist) of knee OA classified K-L Grade 2, 3, or 4 on standing anterior-posterior X-ray of the index knee.
* Osteoarthritis pain in the index knee unresponsive (ie, the participant still experiences pain) to conservative therapy for ≥ 6 months preceding Screening, defined as history indicating that:

  1. Acetaminophen/paracetamol therapy has not provided sufficient pain relief or participant is unable to take acetaminophen/paracetamol chronically/long term because of contraindication or inability to tolerate; AND
  2. At least 1 oral non-steroidal anti-inflammatory drug (NSAID, including cyclooxygenase-2 inhibitors) and/or topical NSAID therapy that has not provided sufficient pain relief or participant is unable to take NSAIDs because of contraindication or inability to tolerate.
* Average WOMAC NRS 3.1 Index pain sub-scale score of 4 to 10 in the index knee at Screening AND a minimum pain score of 4 on either of the individual WOMAC NRS 3.1 Index questions of pain on walking on a flat surface or pain on climbing stairs at Screening.
* Average WOMAC NRS 3.1 Index function sub-scale score of 4 to 10 in the index knee at Screening.
* Body mass index of >=18 to <=39.0 kg/m2
* Female subjects of childbearing potential and Male subjects must agree to comply with protocol specified contraceptive requirements
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Current non-pharmacologic treatment regimen for knee OA (excluding knee brace) must be stable for at least 2 weeks before Day 1 and remain stable throughout the study. Participant must be willing to abstain from starting a new or changing their non-pharmacologic treatment regimen for the duration of the study.
* Willing to stop treatment with oral and topical NSAIDs, and all other systemic pain medications (except acetaminophen/paracetamol per rescue protocol) from 2 weeks before Day 1 to end of study.
* Agrees to use acetaminophen/paracetamol or topical analgesics (topical NSAIDs are prohibited) as rescue therapy if required.

Exclusion Criteria:

* Documented or reported history of increased bleeding in the absence of anticoagulant or antiplatelet drugs or prior history of major bleeding episode in the presence of anticoagulant or antiplatelet therapy.
* History of idiopathic or immune-mediated thrombocytopenia including history of or laboratory confirmed HIT (positive or equivocal antibodies against platelet factor 4 [ie, PF4] and positive Serotonin Release Assay (SRA)].
* Currently active or recent history (within preceding 12 months) of a gastric or duodenal ulcer, or suspicion of gastrointestinal tract bleeding.
* History of other bleeding disorders including haemophilia

  •. Recent cerebral bleeding or operation on brain, spine, or eyes within 6 months of Day 1.
* Spinal anaesthesia within 14 days of Day 1,
* Fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy, or other moderate to severe pain that may confound assessments or self-evaluation of the pain associated with osteoarthritis. Participants with a present (current) history of sciatica are not eligible for participation. Participants with a history of sciatica who have been asymptomatic for ≥ 3 months and who have no evidence of radiculopathy or sciatic neuropathy on thorough neurologic examination are eligible for participation.
* History of other disease that may involve the index joint, including inflammatory joint disease such as rheumatoid arthritis, seronegative spondyloarthropathy (eg, ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease-related arthropathy), crystalline disease (eg, gout), endocrinopathies, metabolic joint diseases, lupus erythematosus, joint infections, Paget's disease, or tumours.
* History of osteonecrosis or osteoporotic fracture (ie, a participant with a history of osteoporosis and a minimally traumatic or atraumatic fracture).
* History of hypersensitivity to PPS, heparin or heparin-like drugs, or drugs of a similar chemical or pharmacological class.
* Predisposition to hypersensitivity due to multiple (2 or more) atopic diseases (such as atopic eczema, asthma, and chronic allergic rhinitis and/or rhinoconjunctivitis) or multiple (2 or more) severe allergies
* Allergy or contraindication to Tetracosactide
* Chronic medical conditions including but not limited to those stated below requiring medical regime changes within 60 days before Day 1. Concurrent unstable peripheral, cardiac, and cerebral vascular disease, poorly controlled chronic obstructive pulmonary disease and asthma, coagulopathies, uncontrolled neurological conditions, active tuberculosis, active infections, symptomatic cardiac arrhythmias, adrenal insufficiency (primary or central), nephrotic syndrome, Cirrhosis (Child-Pugh stage B or C), uncontrolled diabetes and uncontrolled hypothyroidism or hyperthyroidism, or mental or emotional disorders that preclude reliable study participation.
* History of pituitary irradiation or recent (within 1 year) history of transsphenoidal surgery
* Any cancer within the previous 5 years, except for basal cell carcinomas.
* Current hyperkalemia and/or hyponatremia.
* History or current autoimmune polyglandular syndromes
* Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
* Current treatment with anticoagulants or antiplatelet drugs, excluding aspirin ≤100 mg/day.
* Previous treatment with PPS in any form.
* Current or recent (within 90 days before Day 1) immunosuppressive or immunomodulatory (with immunosuppressive effects) systemic therapy including but not limited to oral, inhaled, intranasal, intra-articular and topical corticosteroids (occasional use of topical, inhaled or intranasal corticosteroids is acceptable).
* Use of opioids within 6 weeks before Day 1.
* Use of bisphosphonates within 12 weeks before Day 1.
* Use of denosumab and iloprost within 12 weeks before Day 1.
* Use of a knee brace on the index knee within 2 weeks before Day 1.
* Systemic steroids administered intravenously, intramuscularly, and orally for OA or other indications within 8 weeks before Day 1.
* Intra-articular injections to the index knee: steroids within 24 weeks; hyaluronic acid or any other intra-articular injections within 24 weeks before Day 1.
* Cannabinoids within 30 days before Day 1.
* Use of vitamins and dietary supplements known to alter haemostasis within 2 weeks before Day 1, including ajoene, birch bark, cayenne, Chinese black tree fungus, cumin, evening primrose oil, feverfew, garlic, ginger, ginkgo biloba, ginseng, grapeseed extract, milk thistle, omega 3 fatty acids, onion extract, St. John's wort, turmeric, vitamins C and E, vitamin K.
* Known exposure to heparin within the last 100 days as determined by history of drug use or history of the following medical conditions or interventions: cardiac bypass surgery or thromboembolic disease
* Treatment with dehydroepiandrosterone sulfates within 6 weeks before Day 1.
* Chronic use of oral glucocorticoid receptor antagonists or cortisol synthesis inhibitors within12 weeks before Day 1.
* Biotin within 72 hours of screening.
* Megestrol Acetate within 6 weeks before Day 1
* Current treatment with any medication that may lead to Maculopathy (see Table 3)
* Any medication that alters sodium and/or potassium levels (see Table Prohibited Therapy)
* Participation in another clinical trial or administration of any IP or experimental product within 24 weeks or 5 half-lives (whichever is longer) before Day 1.
* Activated partial thromboplastin time [aPTT]) > 36 seconds, platelets <150,000/µL, or liver enzyme tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) ≥ 2 × ULN at Screening.
* Active or chronic hepatitis B virus, hepatitis C virus, or uncontrolled HIV infection (detectable virus or diagnosis of AIDS); participants with HIV infection must be on chronic suppressive antiviral medication.
* Radiographic evidence of any of the following conditions in any Screening radiograph: excessive malalignment of the knee, severe chondrocalcinosis; other arthropathies (eg, rheumatoid arthritis, psoriatic arthritis, gout), systemic metabolic bone disease (eg, Paget's disease, metastatic calcifications), primary or metastatic tumour lesions, stress, or traumatic fracture.
* Radiographic evidence of any of the following conditions at Screening:

  1. subchondral insufficiency fractures
  2. spontaneous osteonecrosis of the knee
  3. osteonecrosis
  4. pathologic fracture
* Any clinically significant abnormalities on clinical chemistry, haematology, urinalysis, physical examination, medical history, 12-lead ECG, or vital signs as judged by the Investigator (at Screening).
* Resting, supine blood pressure (BP) ≥160 mmHg in systolic pressure or ≥100 mmHg in diastolic pressure at Screening. If a participant is found to have uncontrolled and/or untreated significant hypertension at Screening and anti-hypertensive treatment is initiated, assessment for study eligibility should be deferred until BP and antihypertensive medication have been stable for at least 1 month. For participants with previously diagnosed hypertension, antihypertensive medications must be stable for at least 1 month before Screening.
* Evidence of pigmentary maculopathy identified by a retinal specialist during Screening.
* Morning Cortisol ≤ 3 µg/dL.
* ACTH <10 pg/ml; Morning Cortisol >3 µg/dL and <10 µg/dL and peak cortisol (by ACTH stimulation test) <18 µg/dL.
* Largely or wholly incapacitated (eg, bedridden or confined to a wheelchair, permitting little or no self-care).
* Major surgery or anticipated surgery during the study.
* Currently hospitalized or any planned hospitalizations during the study.
* Plan for total knee reconstruction in affected knee(s) during the study.
* Knee surgery or trauma to the index knee within 1 year before Day 1.
* A history of drug or alcohol abuse and/or dependence within the 12 months before Screening that, in the opinion of the investigator, may affect participant ability to comply with study requirements.
* An employee of the Sponsor, clinical research organisations or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at Day 56 in knee pain as assessed by the average pain sub-scale score of the WOMAC® NRS 3.1 Index. | Baseline, Day 56
  WOMAC: The WOMAC® NRS 3.1 Index is a validated, self-administered, health status questionnaire that assesses pain, stiffness, and function in patients with hip or knee OA . The WOMAC pain sub-scale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee) during the past 48 hours. It is calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS). Scores for each question and WOMAC Pain sub-scale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain.

SECONDARY OUTCOMES:
Key secondary: Change from baseline at Day 56 in function as assessed by the average functional subscale score of the WOMAC NRS 3.1 Index | Baseline to Day 56
  WOMAC: Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function sub-scale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee) during the past 48 hours.
Key secondary: Change from baseline at Day 84 in knee pain as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index | Baseline to Day 84
  WOMAC: The WOMAC pain sub-scale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee) during the past 48 hours.
Key secondary: Change from baseline at Day 84 in function as assessed by the average functional subscale score of the WOMAC NRS 3.1 Index | Baseline to Day 84
  WOMAC: Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function sub-scale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee) during the past 48 hours.
Stage 1 only: Change from baseline at Day 56 and 84 in knee pain as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index for PPS 1.5 mg/kg twice weekly, PPS 2.0mg/kg once weekly, and PPS fixed dose once weekly | Baseline to Day 56 and Day 84
  WOMAC: The WOMAC pain sub-scale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee) during the past 48 hours.
Stage 1 only: Reduction in knee pain of ≥ 30% and ≥ 50% as assessed by the average pain subscale score of the WOMAC NRS 3.1 Index at Days 56 and 84 for PPS 1.5mg/kg twice weekly, PPS 2.0mg/kg once weekly, and PPS fixed dose once weekly | Baseline to Day 56 and Day 84
  WOMAC: The WOMAC pain sub-scale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee) during the past 48 hours.
Stage 1 only: Stage 1 only: Change from baseline at Day 56 and 84 in function as assessed by the average functional subscale score of the WOMAC NRS 3.1 Index for PPS 1.5 mg/kg twice weekly, PPS 2.0mg/kg once weekly, and PPS fixed dose once weekly | Baseline to Day 56 and Day 84
  WOMAC: Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function sub-scale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee) during the past 48 hours.
Stage 1 only: Improvement in function of ≥ 30% and ≥ 50% as assessed by the average functional subscale score of the WOMAC NRS 3.1 Index at Days 56 and 84 for PPS 1.5mg/kg twice weekly, PPS 2.0mg/kg once weekly, and PPS fixed dose once weekly | Baseline to Day 56 and Day 84
  WOMAC: Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function sub-scale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee) during the past 48 hours.
Stage 1 only: PGIC scores at Days 56 and 84 for PPS 1.5mg/kg twice weekly, PPS 2.0mg/kg once weekly, and PPS fixed dose once weekly | Baseline to Day 56 and Day 84
  The PGIC is a self-administered question that rates participants overall improvement in chronic pain since beginning treatment from 1 "no change (or condition has worsened)" to 7 "a great deal better" in response to the question "Since beginning treatment, how would you describe the change (if any) in activity, limitation, symptoms, emotions, and overall QoL related to your arthritis".
Stage 1 and 2: Outcomes Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index response rate at Days 39, 56, 84, 112, 140, and 168 | Baseline, Days 39, 56, 84, 112, 140 and 168
  Participants are considered as an OMERACT-OARSI responder: if the change (improvement) from baseline to day of interest was greater than or equal to >= 50 percent and >= 2 units in either WOMAC pain sub-scale or physical function sub-scale score; if change (improvement) from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain sub-scale score, 2) WOMAC physical function sub-scale score, 3) Patient Global Impression of Change (PGIC).
Stage 1 and 2: Change from baseline at Days 11, 25, 39, 112, 140 and 168 in knee pain as assessed by the average pain sub-scale score of the WOMAC® NRS 3.1 Index. | Baseline, Days 11, 25, 39, 112, 140 and 168
  WOMAC: The WOMAC pain sub-scale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee) during the past 48 hours.
Stage 1 and 2: Change from baseline in knee pain of >=30% and >=50% as assessed by the average pain sub-scale score of the WOMAC® NRS 3.1 Index at Days 11, 25, 39, 112, 140, and 168 | Baseline, Days 11, 25, 39, 112, 140 and 168
  Percentage of participants with reduction in WOMAC pain intensity of at least >=30% or >=50% compared to baseline as assessed by the average pain sub-scale score of the WOMAC® NRS 3.1 Index at Days 11, 25, 39, 56, 84, 112, 140, and 168.
Stage 1 and 2: Change from baseline at Days 11, 25, 39, 112, 140 and 168 in function as assessed by the average functional sub-scale score of the WOMAC® Index. | Baseline, Days 11, 25, 39, 112, 140 and 168
  WOMAC: Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function sub-scale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee) during the past 48 hours.
Stage 1 and 2: Improvement in function of >=30% and >=50% as assessed by the average functional sub-scale score of the WOMAC® NRS 3.1 Index from baseline at Days 11, 25, 39, 112, 140, and 168 | Baseline, Days 11, 25, 39, 112, 140, and 168
  Percentage of participants with improvement in WOMAC function of at least >=30% or >=50% compared to baseline as assessed by the average function sub-scale score of the WOMAC® NRS 3.1 Index at Days 11, 25, 39, 56, 84, 112, 140, and 168.
Stage 1 and 2: Change from baseline at Days 11, 25, 39, 56, 84, 112, 140, and 168 in knee stiffness as assessed by the average stiffness sub-scale score of the WOMAC® NRS 3.1 Index | Baseline, Days 11, 25, 39, 56, 84, 112, 140, and 168
  WOMAC: The WOMAC stiffness sub-scale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the index joint (knee) during the past 48 hours.
Stage 1 and 2: Change from baseline at Days 11, 25, 39, 56, 84, 112, 140, and 168 overall as assessed by the overall score of WOMAC® NRS 3.1 Index | Baseline, Days 11, 25, 39, 56, 84, 112, 140, and 168
  WOMAC: The WOMAC® NRS 3.1 Index consists of 24 questions and produces 3 sub-scales scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarizes overall disability.
Stage 1 and 2: Change from baseline at Days 11, 25, 39, 56, 84, 112, 140, and 168 in Quality of Life (QoL) as assessed by Short Form-36 General Health Survey (SF-36) | Baseline, Days 11, 25, 39, 56, 84, 112, 140, and 168
  The SF-36 v2 is a 36-item, patient-reported survey of patient health, consisting of 8 scaled scores, which are the weighted sums of the questions in their section. The 1-week recall form asks the respondent to answer the questions as they pertain to the way he or she felt or acted during the past week.
Stage 1 and 2: PGIC scores at Days 39, 112, 140, and 168 | Baseline, Days 39, 112, 140, and 168
  The PGIC is a self-administered question that rates participants overall improvement in chronic pain since beginning treatment from 1 "no change (or condition has worsened)" to 7 "a great deal better" in response to the question "Since beginning treatment, how would you describe the change (if any) in activity, limitation, symptoms, emotions, and overall QoL related to your arthritis".
Stage 1 and 2: Change from baseline at Days 56, 84, 112, 140, and 168 in Work Productivity and Activity Impairment (WPAI) questionnaire score | Baseline, Day 56, 84, 112, 140 and 168
  This WPAI questionnaire (WPAI:OA-knee) is a validated self-administered questionnaire that assesses work impairment due to OA . The questionnaire gathers information on employment status, hours worked, hours missed due to OA, and hours missed for any other reasons.
Stage 1 and 2: Number of days of rescue medication used from Day 1 to Day 168 | Baseline up to Day 168
  In case of inadequate pain relief, either acetaminophen/paracetamol up to 3000 mg per day or topical analgesics, up to 4 days in a week could be taken as rescue medication between day 1 and Day 168. Number of participants with any use of rescue medication during the particular study week will be summarized
Stage 1 and 2: Incidence of treatment-emergent Adverse Event (TEAEs), including serious AEs (SAEs) | Baseline up to Day 168
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
  An SAE is any untoward medical occurrence that at any dose results in one or more of the following outcomes: death; life-threatening; requires in-patient hospitalization or prolongation of an existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; is an important medical event. Treatment-emergent are events between the first dose of study drug and up to Day 168 that were absent before treatment or that worsened relative to pre-treatment state.
Stage 1 and 2: Treatment-emergent clinical laboratory abnormalities | Baseline up to Day 168
  Treatment-emergent clinical laboratory abnormalities are abnormalities in labs between the first dose of study drug and up to Day 168 that were absent before treatment or that worsened relative to pre-treatment state
Stage 1 and 2: Clinically significant changes in electrocardiograms (ECG) compared with baseline (pharmacokinetic [PK] subset only) | Baseline, Day 1, Day 15, Day 36 and Day 39
  Clinically significant changes in ECGs between the first administration of study drug and up to Day 39 that were absent before treatment or that worsened relative to pre-treatment state.

OTHER OUTCOMES:
Exporatory: Number of participants with an Anti-Drug-Antibody (ADA) response after treatment | Baseline, Days 11, 25, 39, 56 and 84
  Human serum ADA samples will be analyzed for the presence or absence of anti-drug-antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA).
Exploratory: Correlation of Anti-Drug-Antibody (ADA) response with clinical events | Baseline, Days 11, 25, 39, 56, and 84
  Human serum ADA samples will be analyzed for the presence or absence of anti-drug-antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA).
Exploratory: PPS PK profile of single and multiple doses based on sparse blood sampling | Stage 1: Day 1, 15 and 39 - pre-dose and 2, 4, and 6 hours. Pre-dose on Days 4, 8, 11, 18, 22, 25, 29, 32 and 36
  Blood samples for assay of plasma PPS concentration will be obtained from a subset of patients before dosing and 2, 4, and 6 hours after dosing on study Days 1,15 and 39, and assayed using a sensitive, validated [binding, etc.] bioanalytical method. Plasma concentrations of PPS will be tabulated by time and participant and inspected for relationship to dose during titration and stable treatment phases.
Exploratory: Change in subchondral BML area and volume on MRI from baseline at Day 168 | screening, Day 168
  Bone Marrow lesions (BML) will be evaluated for changes based on MRI imaging
Exploratory: The effect of PPS on subchondral BML volume and area on MRI and whether these changes correlate with clinical outcomes | screening, Day 168
  Bone Marrow lesions (BML) will be evaluated for changes based on MRI imaging
Exploratory: Changes in joint synovitis/effusion volume on MRI from baseline on Day 168 | screening, Day 168
  Synovitis/effusion will be evaluated for changes based on MRI imaging
Exploratory: The effect of PPS on joint synovitis/effusion volume on MRI and whether these correlate with clinical outcomes | screening, Day 168
  Synovitis/effusion will be evaluated for changes based on MRI imaging
Exploratory: Change in cartilage volume on MRI from baseline at Day 168 | screening, Day 168
  Cartilage volume will be evaluated for changes based on MRI imaging
Exploratory: The effect of PPS on cartilage volume changes on MRI and whether these correlate with clinical outcomes | screening, Day 168
  Cartilage volume will be evaluated for changes based on MRI imaging
Exploratory: Change in bone shape on MRI from baseline at Day 168 | screening, Day 168
  Bone shape will be evaluated for changes based on MRI imaging
Exploratory: The effect of PPS on bone shape changes and whether these correlate with clinical outcomes | screening, Day 168
  Bone shape will be evaluated for changes based on MRI imaging
Exploratory: Change in joint space width on MRI from baseline at Day 168 | screening, Day 168
  Joint space will be evaluated for changes based on MRI imaging
Exploratory: The effect of PPS on joint space width changes and whether these correlate with clinical outcomes | screening, Day 168
  Joint space will be evaluated for changes based on MRI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schnitzer, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (33):
- United States (29):
  - Alliance for Multispecialty Research - Tempe, Tempe, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Core Healthcare Group, Cerritos, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Providence Clinical Research, North Hollywood, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Encompass Clinical Research, Spring Valley, California
  - Clinical Research of West Florida- Clearwater, Clearwater, Florida
  - University Clinical Research-Deland, DeLand, Florida
  - LMG Research, Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Alliance for Multispecialty Research - Newton, Newton, Kansas
  - Alliance for Multispecialty Research - Wichita West, Wichita, Kansas
  - Alliance for Multispecialty Research - Wichita East, Wichita, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Alliance for Multispecialty Research - Las Vegas, Las Vegas, Nevada
  - Kaplan Medical Research, Las Vegas, Nevada
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Alliance for Multispecialty Research - Knoxville, Knoxville, Tennessee
  - FutureSearch Trials - Austin, Austin, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Diagnostics Research Group - Northwest San Antonio, San Antonio, Texas
  - Discovery Clinical Trials, San Antonio, Texas
- Australia (4):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Griffith University, Southport, Queensland
  - Sportsmed, Stepney, South Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No